CLINICAL TRIAL: NCT04185701
Title: Study of the Subjective Refraction Measured With SiVIEW Software Compared to That Obtained Manually by an Expert. Monocentric Cross-sectional Study
Brief Title: Comparison of Subjective Refraction Measurement With SiVIEW Software and by an Expert
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SiVIEW (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: SiVIEW_refraction_Paris_study
Record Dates: First submitted 2019-11-30; First posted 2019-12-04 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-03

CONDITIONS: Eye Diseases; Ametropia
Keywords: automatic sphere measurements; eye examination; ametropia
MeSH Terms: conditions — Eye Diseases; Refractive Errors

STUDY DESIGN:
Intervention Model Description: * Eye examination by an expert including optimal correction in distance and near vision
  * Eye examination by a technician with the SiVIEW system
  * Analysis of the SiVIEW report by the expert who conducted the second review
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eye examination by expert and SiVIEW software (Experimental): Eye examination by an expert and by a technician with the SiVIEW system.
  Interventions: Other: SiVIEW software; Other: Expert

INTERVENTIONS:
Other: SiVIEW software — Eye examination by a technician with the SiVIEW software
Other: Expert — Eye examination by an expert including optimal correction in distance and near vision

SUMMARY:
Main objective

Show that the equivalent sphere refraction measurements obtained by the SiVIEW software have no significant clinical difference with those obtained by an optometrist expert.

Secondary objectives

Show that the sphere refraction measurements obtained by the SiVIEW software have no significant clinical difference with those obtained by an optometrist expert.

Show that the cylinder refraction measurements obtained by the SiVIEW software have no significant clinical difference with those obtained by an optometrist expert.

Show that the visual acuity measurements obtained by the SiVIEW software do not have a significant clinical difference with those obtained by an optometrist expert.

Demonstrate that the report delivered for each eye exam by SiVIEW software is consistent and relevant to a vision health practitioner.

Show that the differences obtained between two eye examination experts are consistent with those found in the literature.

DETAILED DESCRIPTION:
Introduction:

Ametropia is an eye refractive disorder typically leading to myopia, hyperopia, astigmatism... 4.5 billion people are currently affected worldwide, of whom only 2 billion are corrected. Of these people, about 30% (or +/- 600,000) do not benefit from an adequate correction. From an economic point of view, the cost on productivity of the absence or poor vision correction is estimated at more than 270 billion euros / year worldwide.

Any correction of an ametropic disorder necessarily requires a precise and relevant eye examination in order to identify the disorder and determine the best possible visual correction. The procedure for this examination is identical in all countries. It must follow specific steps[Benjamin 2006; Grosvenor 2007].

At present the refraction measurement is done manually by an expert. The optical correction may vary from one examination to another, for multiple physiological and/or examination-related reasons. Several factors can cause fluctuations in subjective refraction. These include examiner and subject characteristics [Grein et al. 2014].

In addition, there is also variability due to the measurement itself, depending on each examiner. The repeatability (on the same subject) and, in addition, the reproducibility (inter-examiners) of the subjective refraction measurement related to the examiner's interpretation, examination process and experience, among other things, are therefore important data to be defined in order to know the tolerance of the measurement determined between two examinations.

In studies involving a large number of subjects, the repeatability/reproducibility limit is greater than or equal to 0.71D [Zadnik 1994, Bullimore 1998, MacKenzie 2008], and more particularly during inter-examiner measurements.

The objective of the SiVIEW solution is therefore to make the measurement of subjective refraction both repeatable and reproducible regardless of the practitioner and his expertise, by completely automating the search for the best visual prescription using an expert system that aims to make this examination simple, intuitive and reliable.

It is therefore essential to compare the SiVIEW measurement with that of an optometrist expert.

The interest of the investigator's study will be to demonstrate that the results between a refraction expert and the measurement obtained by SiVIEW are clinically similar.

Main objective:

Show that the equivalent sphere refraction measurements obtained by the SiVIEW software have no significant clinical difference with those obtained by an optometrist expert.

Secondary objectives

Show that the sphere refraction measurements obtained by the SiVIEW software have no significant clinical difference with those obtained by an optometrist expert.

Show that the cylinder refraction measurements obtained by the SiVIEW software have no significant clinical difference with those obtained by an optometrist expert.

Show that the visual acuity measurements obtained by the SiVIEW software do not have a significant clinical difference with those obtained by an optometrist expert.

Demonstrate that the report delivered for each eye exam by SiVIEW software is consistent and relevant to a vision health practitioner.

Show that the differences obtained between two eye examination experts are consistent with those found in the literature.

Plan of the study:

It is a comparative prospective open monocentric cross-sectionnal study.

ELIGIBILITY:
Inclusion Criteria:

* subject with visual AV on each eye >= 8/10 and no amblyopia
* subject with normal environmental transparency
* subject with a healthy fundus that does not reveal major abnormalities that may affect vision
* subject able to read the letters of the Latin alphabet
* subject without heavy drug treatment that may affect vision as synthetic antimalarials, corticosteroids
* non-diabetic subject
* non nystagmic subject
* non-strabic subject
* subject who has not had eye surgery less than 1 year old

Exclusion Criteria:

* subject with a topography showing an anomaly (keratoconus type or other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Equivalent sphere measurement | At time of inclusion
  The subject will have an eye exam with SiVIEW and an examination by an optometrist expert. The equivalent sphere value will be evaluated in both cases.

SECONDARY OUTCOMES:
Sphere measurement | At time of inclusion
  The subject will have an eye exam performed with SiVIEW and by an optometrist expert. The sphere value will be evaluated in both cases. The examination will be started in both cases on the objective measurement value obtained during the routine care examination.
Cylinder measurement | At time of inclusion
  The subject will have an eye exam performed with SiVIEW and by an optometrist expert. The cylinder value will be evaluated in both cases. The examination will be started in both cases on the objective measurement value obtained during the routine care examination.
Visual acuity | At time of inclusion
  The subject will have an eye exam performed with SiVIEW and by an optometrist expert. The value of visual acuity will be assessed in both cases.
Consistency and relevance of the SiVIEW report | At time of inclusion
  After each examination, the report edited by the SiVIEW software will be scored consistently on a Likert scale from 1 to 5 by an expert optometrist:
  1: very inconsistent / 2: inconsistent / 3: no opinion / 4: consistent / 5: very consistent
  After each examination, the report edited by SiVIEW software will be scored in relevance on a 5 item Likert scale by an expert optometrist:
  1: not relevant / not very relevant / no opinion / relevant / very relevant.
Measurement between two optometrist experts | At time of inclusion
  Each subject will have an eye examination conducted with an optometrist from the current care centre and by an optometrist expert mandated by SiVIEW (who is used to working at the Rothschild Foundation in clinical studies, among others). The equivalent sphere value will be evaluated in both cases.

CONTACTS AND LOCATIONS:
Overall Officials: Damien Gatinel, MD, Principal Investigator — Head of Department Ophthalmological Foundation A. de Rothschild, Paris, France
Locations (1):
- Ophthalmological Foundation A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No